CLINICAL TRIAL: NCT06828991
Title: ctDNA-Guided Mosunetuzumab Consolidation Therapy in Older Patients With Untreated DLBCL
Brief Title: A Study to Evaluate the Impact of Mosunetuzumab Consolidation for Older Patients With Diffuse Large B-cell Lymphoma (DLBCL) Who Have Detectable Amounts of ctDNA (Circulating Tumor DNA) at the End of Treatment With Pola-R-mini-CHP
Acronym: GOLD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Danielle Wallace (Other)
Collaborators: Genentech, Inc. (Industry); Adaptive Biotechnologies (Industry); Lymphoma Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Danielle Wallace, Assistant Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMLYM24067
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: Diffuse large B-cell lymphoma; Mosunetuzumab; circulating tumor DNA; Measurable residual disease; Geriatric assessment
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Single center, open-label, single arm, phase II pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ctDNA positive (Experimental): Patients who have achieved a radiographic complete response (CR) on PET/CT, but have detectable ctDNA at the end of treatment with pola-R-mini-CHP will receive 6 cycles of mosunetuzumab consolidation. Patients who have achieved a CR with undetectable ctDNA will be observed. Patients with a partial response on PET/CT will be managed per protocol.
  Interventions: Drug: Mosunetuzumab; Device: ClonoSEQ

INTERVENTIONS:
Drug: Mosunetuzumab — Mosunetuzumab consolidation therapy will consist of 6 cycles of IV mosunetuzumab at the standard ramp-up dosing (Day 1 1mg, Day 8 2mg, D15 60mg, C2D1 60mg, and 30mg on day 1 of the subsequent 21-day cycles)
  Other Names: Lunsumio
Device: ClonoSEQ — Patients with detectable ClonoSEQ at C6D1 who have a PET/CT that shows a CR will receive mosunetuzumab

SUMMARY:
Older patients with diffuse large B- cell lymphoma (DLBCL) do not have the same rates of disease control as younger patients and are at risk for toxicity. Identifying which patients might benefit from more therapy at the end of first-line treatment is important. The ability to measure small amounts of persistent lymphoma (circulating tumor DNA or ctDNA) might allow the investigators to risk stratify patients. If older patients have detectable ctDNA in the blood at the end of six cycles of polatuzumab vedotin, rituximab and dose-attentuated CHP chemotherapy, patients will receive a bispecific antibody called mosunetuzumab. The investigators hypothesize this will result in "clearing" the ctDNA from the blood and result in better disease control and outcomes for patients. The study will also measure the safety of this regimen and the impact on the function of these older patients utilizing a tool called the geriatric assessment.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged greater than or equal to 70 years of age who are ineligible for full-intensity chemoimmunotherapy at the discretion of the treating investigator. If between the ages of 70-79, the reason for ineligibility should be documented in a clinical note. If 80 or older, the reason for dose-attenuated chemoimmunotherapy is assumed to be age.
2. ECOG performance status of 0-2.
3. Histologically-confirmed DLBCL, NOS, high grade B-cell lymphoma with MYC and BCL2 rearrangements, high grade B-cell lymphoma, NOS, and grade 3b follicular lymphoma
4. Histologic transformation (HT) will be included on the study. This must be confirmed with a biopsy. Patients with HT may have received prior treatment for indolent lymphoma including chemoimmunotherapy but must not have received an anthracycline-containing regimen in the past.
5. Composite and discordant lymphomas containing both indolent and large cell features will be included.
6. Has received no prior therapy for aggressive B-cell lymphoma or HT with the following exceptions: a course of corticosteroids given for lymphoma related symptoms or one cycle of anthracycline containing chemotherapy prior to enrollment on the clinical trial. Pre-phase treatment with polatuzumab vedotin and steroids is allowable at the treating investigator's discretion.
7. Ejection fraction of ≥ 45% on echocardiogram or MUGA
8. Patient has a platelet count of ≥75,000/µL within the screening period unless inadequate function is due to bone marrow infiltration with aggressive B-cell lymphoma in which case the platelet count should be ≥ 30,000/µL
9. Patient has an absolute neutrophil count of ≥1,500/ µL within the screening period unless inadequate function is due to bone marrow infiltration with aggressive B-cell lymphoma in which case the neutrophil count should be ≥500/ µL
10. Patient has a calculated or measured creatinine clearance of >40 mL/minute within the screening period.
11. Total bilirubin must be less than 1.5 times the upper limit of normal (ULN) unless the elevation is known to be due to Gilbert syndrome or hepatic involvement with aggressive B-cell lymphoma in which case it can be ≤ 3.0 times the ULN. ALT or AST must be ≤ 2.5 times the ULN.
12. Patient has, with treatment in the opinion of the treating investigator, a life expectancy of at least 12 weeks.
13. Signed Informed Consent Form
14. Ability to comply with the study protocol

Exclusion Criteria

Patients who meet any of the following exclusion criteria are not to be enrolled to this study:

1. History of, or clinically apparent central nervous system (CNS) lymphoma
2. Primary mediastinal B-cell lymphoma
3. Patient is receiving peritoneal dialysis or hemodialysis
4. Patient has > Grade 1 peripheral neuropathy.
5. EF <45% or significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 6 months prior to the start of Cycle 1, unstable arrhythmias, or unstable angina
6. Patient has received other investigational drugs within 28 days before enrollment.
7. Prior exposure to anthracycline
8. Patient has concomitant active malignancy that the treating physician or PI feels may interfere with the ability to measure the primary or secondary outcomes. Patients with stage 1 cancers are eligible after definitive treatment. Patients with low grade prostate cancer who are managed with observation are eligible. Patients with other malignancies that have been treated with curative intent may be included after discussion with the study PI.
9. Participants who have a positive HIV test at screening, with the following exception: Individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy for at least 4 weeks, have a CD4 count >/= 200/uL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months.
10. Patient has active hepatitis B with a positive surface antigen or viral load. Carriers of hepatitis B virus should be closely monitored for clinical and laboratory signs of active HBV infection and for signs of hepatitis throughout study participation according to national and local guidelines. Those at high risk of reactivation should be placed on appropriate antiviral therapy as per national guidelines.
11. History of solid organ transplantation, or post-transplant lymphoproliferative disorder.
12. Patient has history of allogeneic stem cell transplantation.
13. Serious medical or psychiatric illness likely to interfere with participation in this clinical study including clinically significant CNS disease, active infections, or autoimmune disease that in the opinion of the treating investigator impacts their ability to safely participate in the clinical trial.
14. Any clinically significant abnormality in screening blood chemistry, hematology, or urinalysis results that, in the judgment of the investigator, would impede adequate evaluation of adverse events and/or response to treatment, or that requires aggressive intervention.
15. Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone (>20 mg), azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents within 2 weeks prior to Day 1 of the first cycle of mosunetuzumab. The use of inhaled corticosteroids is permitted, as is the use of mineralocorticoids for management of orthostatic hypotension and a dose of dexamethasone 20mg or less for nausea or B symptoms.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance rate after mosunetuzumab treatment | From the beginning to the end of mosunetuzumab treatment at 18 weeks
  The primary endpoint of the trial is the ctDNA clearance rate after mosunetuzumab treatment among the subset of patients in a PET/CT CR but with ctDNA+ at the end of 6 cycles of R-pola-mini-CHP. The rate will be calculated as the number of subjects ctDNA- after mosunetuzumab treatment among all patients treated with mosunetuzumab as part of the Fleming two-stage design.

SECONDARY OUTCOMES:
Objective response rate and complete response rate of pola-R-mini-CHP | From enrollment to the end of pola-R-mini-CHP treatment at 18 weeks
  Objective response rate is the number of patients in the study population who achieve a complete or partial response to therapy, the complete response rate is only those patients who achieve a complete response.

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At time of publication
Access Criteria: At request of other researchers at time of publication